CLINICAL TRIAL: NCT06528743
Title: Feasibility of Primer Shot Radiotherapy for Non-small Cell Lung Cancer - PRIMER
Acronym: PRIMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: N23PSR
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Patients With Non-small-cell Lung Cancer

STUDY DESIGN:
Intervention Model Description: Initially, patients are included following a 3+3 design to find the maximum tolerated break length, followed by an expansion cohort (unless there are already 2+ patients drop out in schedule 1, then there will be no expansion cohort).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primer shot treatment break of 1 week (Experimental): Patients receive an increasing primer shot treatment break. In arm 1, the break between the first and the second radiotherapy fraction is 1 week
  Interventions: Radiation: RT (5x6 Gy) to the primary tumor and, if indicated, to lymph node and/or distant metastases.
- Primer shot treatment break of 2 weeks (Experimental): Patients receive an increasing primer shot treatment break. In arm 1, the break between the first and the second radiotherapy fraction is 2 weeks
  Interventions: Radiation: RT (5x6 Gy) to the primary tumor and, if indicated, to lymph node and/or distant metastases.
- Primer shot treatment break of 3 weeks (Experimental): Patients receive an increasing primer shot treatment break. In arm 1, the break between the first and the second radiotherapy fraction is 3 weeks
  Interventions: Radiation: RT (5x6 Gy) to the primary tumor and, if indicated, to lymph node and/or distant metastases.

INTERVENTIONS:
Radiation: RT (5x6 Gy) to the primary tumor and, if indicated, to lymph node and/or distant metastases. — Patients will receive RT (5x6 Gy) to the primary tumor and, if indicated, to lymph node and/or distant metastases. Enrolled patients will receive a fractionation scheme with increasing break length.

SUMMARY:
Intro/rationale: Radiotherapy employs uniform, equally spaced weekday fractions that do not account for changes in tumor radiosensitivity. However, radiobiological characteristics evolve during the radiotherapy schedule as reoxygenation increases radiosensitivity. In tumor-response simulations and preclinical experiments, it was superior to prime the tumor with one radiotherapy fraction, followed by a treatment break permitting mitotic cell death and reoxygenation of tumor cells.

Objective: To determine the safety and feasibility of primer shot fractionation for NSCLC.

Study design: A prospective non-randomized feasibility trial to test the safety of primer shot fractionation in a 3+3 phase with increasing treatment breaks, followed by an expansion cohort.

Study population: Patients with NSCLC stage 2-4, referred for palliative radiotherapy of the primary tumor and possibly (lymph node) metastases. Patients are allowed to receive systemic treatments, except for VEGFR-inhibitors. The 3+3 phase is followed by an expansion phase of 22 patients.

Intervention: All treatments are 5x6 Gy to all targets. Patients receive an increasing primer shot treatment break. In the 3+3 phase, the break between the first and the second radiotherapy fraction is: 1, 2 and 3 weeks. The maximum tolerated break length will be used for the expansion cohort.

Main study parameters/endpoints: The main study endpoint is the ability of patients to finish the radiotherapy schedule as planned. Secondary endpoints are tumor response at the end of treatment and 3 months thereafter, and acute toxicity.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Based on simulations and preclinical data, primer shot treatment breaks increase tumor control. However, the increased overall treatment time could potentially increase the chance a patient drops out before the radiotherapy schedule is finished. Because of the gradually prolonged break, this risk is relatively small and acceptable for this population. Additionally, patients are asked to fill in PRO-CTCAE lung subset questionnaires at the start of treatment and during follow-up. They will also receive 1 additional CT with contrast at fraction 5.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* NSCLC (either pathology proven or sufficient clinical suspicion to be treated as NSCLC), referred for palliative radiotherapy of at least the primary tumor site.
* Stage 2-4
* WHO performance score 0-2.
* Provision of signed, written and dated IC prior to any study specific procedures.

Exclusion Criteria:

* Interstitial lung disease
* Treatment with vascular endothelial growth factor receptor (VEGFR) inhibitors
* Prior thoracic radiotherapy (>20 Gy EQD2 a/b 3) overlapping with the current planning target volume

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
the ability of patients to finish the radiotherapy schedule | 5 weeks
  The study is powered to find a decrease of response from 99% to no less than 84.15% (relative decrease of 15%).

SECONDARY OUTCOMES:
Tumor response | at the end of treatment and after 3 months
  the relative volume change after radiotherapy vs the CTRT.
treatment associated ≥ grade 2 non-hematologic toxicity according to the NCI Common Terminology Criteria of Adverse Events (CTCAE version 5.0) (from the first radiotherapy fraction until 6 months after radiotherapy) | from the first radiotherapy fraction until 6 months after radiotherapy
Patient-reported outcome patient-reported outcome- Common Terminology Criteria of Adverse Events (PRO)-CTCAE | up to 1 year after radiation.

CONTACTS AND LOCATIONS:
Locations (1):
- Het Nederlands Kanker Instituut-Antoni van Leeuwenhoek Ziekenhuis Stichting, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided